CLINICAL TRIAL: NCT00606138
Title: Investigation of Ranibizumab for the Treatment of Persistent Diabetic Neovascularization as Assessed by Super Wide-Field Angiography (Optos)
Brief Title: Ranibizumab for Treatment of Persistent Diabetic Neovascularization Assessed by Wide-Field Imaging
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 06120402
Record Dates: First submitted 2008-01-09; First posted 2008-02-01 (Estimated); Results first posted 2014-11-06 (Estimated); Last update posted 2023-04-10 (Actual); Status verified 2023-04

CONDITIONS: Proliferative Diabetic Retinopathy
MeSH Terms: interventions — Ranibizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Anti-VEGF injection (Experimental): Intravitreal injection of 0.5-mg dose of ranibizumab
  Interventions: Drug: ranibizumab
- PRP Laser (Active Comparator): Additional panretinal photocoagulation (up to 500 300-500 um laser spots)
  Interventions: Procedure: Laser photocoagulation

INTERVENTIONS:
Drug: ranibizumab — One 0.5 mg intravitreal injection
  Other Names: Lucentis
  Arms: Anti-VEGF injection
Procedure: Laser photocoagulation — panretinal photocoagulation (up to 500 300-500 um laser spots)
  Arms: PRP Laser

SUMMARY:
Diabetic neovascularization refers to a type of diabetic retinopathy which is worsening by the abnormal growth of blood vessels in the back of the eye, damaging the retina. The usual treatment is a type of laser, called panretinal photocoagulation. One drawback is that the amount of space within the eye for use of this treatment eventually has its limit, and should not be used too near the part of the retina used for detailed vision (the macula). In similar eye disorders, there are certain injectable medications called anti-VEGF treatments which can slow down or stop this abnormal blood vessel growth. This study sought to compare use of ranibizumab versus standard panretinal photocoagulation in treatment of diabetic neovascularization.

DETAILED DESCRIPTION:
The purpose is to compare the efficacy of ranibizumab versus additional panretinal photocoagulation on diabetic neovascularization that is persistent despite previous treatment with panretinal photocoagulation. We hypothesize that ranibizumab intravitreal injections would induce neovascular regression in similar or better fashion than supplemental laser photocoagulation. Consented, enrolled subjects will either receive open-label intravitreal injections of 0.5-mg dose of ranibizumab or additional panretinal photocoagulation (up to 500 300-500 um laser spots) in a ratio of two-to-one (2:1) at the beginning of the study period. ETDRS best-corrected visual acuity, contrast sensitivity, and Optos color photography will be performed at enrollment, at weeks 1, 2, 3 and 4, and at months 2, 3, 4, 5 and 6. The subjects will undergo fluorescein angiography utilizing the Optomap FA (fluorescein angiography) system and optical coherence tomography (OCT) at enrollment, at weeks 2 and 4, and at months 2, 3, 4 and 6. The subjects will be followed for a 6-month period for stabilization, regression, or recurrence of neovascularization. In addition, patients will be evaluated for occurrence of macular edema.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide written informed consent and comply with study assessments for the full duration of the study
* Age 18 years or older

Patient related considerations:

* Patients with Diabetes Mellitus (Type I or II) are eligible. HgA1c will be evaluated at the beginning of the study, but this value will have no significance in inclusion or exclusion.
* Patients will not be pregnant at enrollment and must provide evidence of the use of two types of birth control while enrolled in the study.
* Patients will have no known sensitivity to ranibizumab or other anti-VEGF injections.

Disease related considerations:

* Patients will have diabetic neovascularization as seen on fluorescein angiography that was previously treated with full (at least 1200 laser burns) panretinal photocoagulation and that has persisted at least three months.
* There will be no evidence of ocular inflammation at enrollment.
* There is no restriction on patient's current medications or concomitant illnesses as long as there is no interference with patient follow-up.

Other considerations:

* Patients may not be enrolled in another clinical study or observational trial.
* There is no limitation on patient's institutional status as long as the patient is able to participate in follow-up.

Exclusion Criteria:

* Pregnancy (positive pregnancy test)
* Uncontrolled glaucoma on three medicines or more to control intraocular pressure
* Prior enrollment in the study
* Any other condition that the investigator believes would pose a significant hazard to the subject if the investigational therapy were initiated
* Participation in another simultaneous medical investigation or trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2008-01; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mathew W MacCumber, MD, PhD, Principal Investigator — Rush University Medical Center
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects will be recruited starting in 2007 and until sufficient subject population is reached. They will be seen in an eye clinic at Rush University Medical Center.
Pre-assignment Details: There is no wash-out period. Recruited subjects must be in need of treatment for their PDR, and will be randomized and treated at the baseline visit. There were a total of 8 participants treated.
Groups:
- 1 - Ranibizumab: Intravitreal injection of 0.5-mg dose of ranibizumab
- 2 - Additional PRP Treatment: Additional panretinal photocoagulation (up to 500 300-500 um laser spots)
Period: Overall Study
Arm/Group | 1 - Ranibizumab | 2 - Additional PRP Treatment
Started | 6 | 2
Completed | 4 | 2
Not Completed | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 1 - Ranibizumab | 2 - Additional PRP Treatment | Total
Number analyzed (Participants) | 6 | 2 | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 1 | 7
  >=65 years | 0 | 1 | 1
Age, Continuous [Median (Full Range); unit: years] | 57 [50 to 62] | 67 [60 to 73] | 59 [50 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 5 | 1 | 6
Region of Enrollment [Number; unit: participants]
  United States | 6 | 2 | 8

OUTCOME MEASURES:

1. Primary Outcome: The Mean Percentage Change of the Area of the Patient's Neovascularization as Measured in Pixels by Optomap FA (Fluorescein Angiography)
Description: This is a measurement of how much change in neovascularization has occurred, using the Optomap FA readings to calculate the increase or decrease in surface area of the retina that is affected by neovascularization.
Time Frame: Baseline to Week 4; Baseline to Month 4-6
Measure: Mean (Standard Deviation); unit: percentage of change in area (mean)
Arm/Group | 1 - Ranibizumab | 2 - Additional PRP Treatment
Number analyzed (Participants) | 6 | 2
percentage of change in area (mean)
  Change at Week 4 from baseline | -83.8 (NA) — Data can't be calculated due to lack of original case reports | 52.6 (NA) — Data can't be calculated due to lack of original case reports
  Change at Month 4-6 from baseline | 11.3 (NA) — Data can't be calculated due to lack of original case reports | 55.4 (NA) — Data can't be calculated due to lack of original case reports

2. Primary Outcome: The Mean Percentage Change of Macular Edema Measured by Retinal Thickness by OCT (Optical Coherence Tomography)
Time Frame: Baseline to Week 4; Baseline to Month 6
Measure: Mean (Standard Deviation); unit: percentage of change (mean)
Arm/Group | 1 - Ranibizumab | 2 - Additional PRP Treatment
Number analyzed (Participants) | 6 | 2
percentage of change (mean)
  Change from Baseline to Week 4 | -2.4 (NA) — Data can't be calculated due to lack of original case reports | -8.4 (NA) — Data can't be calculated due to lack of original case reports
  Change from baseline to Month 6 | 54.1 (NA) — Data can't be calculated due to lack of original case reports | -2.1 (NA) — Data can't be calculated due to lack of original case reports

3. Primary Outcome: Incidence and Severity of Ocular Adverse Events, as Identified by Ophthalmic Examination
Time Frame: Month 6
Measure: Number; unit: number of events
Arm/Group | 1 - Ranibizumab | 2 - Additional PRP Treatment
Number analyzed (Participants) | 6 | 2
number of events | 0 | 1

4. Primary Outcome: Number of Participants With Occurrence of Adverse Events
Description: Patients were randomized to receive IVR vs. additional PRP. Number of participants with adverse events.
Time Frame: Week 1, 2, 4; Month 2, 3, 4, 5, 6
Measure: Count of Participants; unit: Participants
Arm/Group | Anti-VEGF Injection | PRP Laser
Number analyzed (Participants) | 6 | 2
Participants | 0 | 2

5. Secondary Outcome: Mean Change in Best Corrected Visual Acuity (BCVA), as Assessed by the Number of Lines Gained on the ETDRS Eye Chart at a Starting Test Distance of 4 Meters
Time Frame: 1 Month; 6 months
Measure: Mean (Standard Deviation); unit: lines of vision gained
Arm/Group | 1 - Ranibizumab | 2 - Additional PRP Treatment
Number analyzed (Participants) | 6 | 2
lines of vision gained
  Week 4 | 2 (1) | 0 (1)
  Month 6 | 3 (1.5) | 2 (1.5)

6. Secondary Outcome: Percentage of Patients Gaining 3 or More Lines of Vision According to ETDRS Eye Chart Testing
Time Frame: 1 month, 6 months
Measure: Number; unit: percentage of participants
Arm/Group | Anti-VEGF Injection | PRP Laser
Number analyzed (Participants) | 4 | 2
percentage of participants
  Percentage of Participants with Lines gained in BCVA at 1 mos | 50.0 | 0
  Percentage of Participants with Lines gained in BCVA at 6 mos | 75.0 | 33.33

7. Secondary Outcome: Occurrence Rate of Proliferative Diabetic Complications Including Vitreous Hemorrhage, Iris Neovascularization, and Tractional Retinal Detachment
Description: Complications; including vitreous hemorrhage, iris neovascularization, and tractional retinal detachment were assessed at the 6 month time point and are reported below.
Time Frame: 6 month
Measure: Number; unit: number of PDR complications
Arm/Group | 1 - Ranibizumab | 2 - Additional PRP Treatment
Number analyzed (Participants) | 6 | 2
number of PDR complications | 0 | 1

ADVERSE EVENTS:
Time Frame: Up to a maximum of 6 months or 14 days after early study withdrawal.
Description: There are no oddities regarding definitions of adverse events for this study nor the collection or reporting thereof.
Arm/Group | 1 - Ranibizumab | 2 - Additional PRP Treatment
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/2
Other Adverse Events (participants affected / at risk) | 0/6 | 2/2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1 - Ranibizumab (N=6) | 2 - Additional PRP Treatment (N=2)
Eye injury, mild, unrelated to treatment (Eye disorders) | 0 (0) | 1 (1) — Subject experienced pain and mild subjconjunctival hemorrhage due to a minor blow to the eye during gardening; unrelated to study participation
Vitreous Hemorrhage (Eye disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2007-08-15): https://cdn.clinicaltrials.gov/large-docs/38/NCT00606138/Prot_000.pdf
  • Informed Consent Form (2010-08-02): https://cdn.clinicaltrials.gov/large-docs/38/NCT00606138/ICF_001.pdf